CLINICAL TRIAL: NCT02029612
Title: An Evidence Based Smoking Cessation Program for Persons Living With HIV/AIDS
Brief Title: An Evidence Based Smoking Cessation Program for Persons Living With HIV/AIDS (Project Legacy)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Centers for Medicare and Medicaid Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2013-0495
Record Dates: First submitted 2013-11-19; First posted 2014-01-08 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Tobacco Use Cessation
Keywords: Tobacco Use Cessation; Cancer Prevention; HIV/AIDS; Questionnaires; Surveys; Nicotine patch; Breath test; Cell Phone Calls for Smoking Cessation Counseling; Text Message Smoking Cessation Support
MeSH Terms: conditions — Tobacco Use Cessation; Acquired Immunodeficiency Syndrome | interventions — Tobacco Use Cessation Devices; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 - Phone Call Support (Other): Smoking cessation telephone hotline phone number provided to participants, along with a 10 week supply of nicotine patches. Each participant counseled on quitting smoking at baseline. Questionnaires completed at baseline, 3 months, and at 6 months. Participant receives 11 phone calls from study staff over a 6-month period. Breath test performed at 3 month and 6 month visit.
  Interventions: Drug: Nicotine Patch; Behavioral: Phone Counseling; Behavioral: Questionnaires; Behavioral: Breath Test; Behavioral: Proactive Cell Phone Smoking Cessation Counseling
- Group 2 - Text Messaging Support (Other): Participants receive 10 week supply of nicotine patches. Each participant counseled on quitting smoking at baseline. Questionnaires completed at baseline, 3 months, and at 6 months. Participants receive text messages for support about quitting smoking over a 6 month period. Breath test performed at 3 month and 6 month visit.
  Interventions: Drug: Nicotine Patch; Behavioral: Phone Counseling; Behavioral: Questionnaires; Behavioral: Breath Test; Behavioral: Text Message Smoking Cessation Support

INTERVENTIONS:
Drug: Nicotine Patch — 10 week supply of nicotine patches given to participants at baseline.
Behavioral: Phone Counseling — Each participant counseled on quitting smoking at baseline.
Behavioral: Questionnaires — Questionnaires completed at baseline, 3 months, and at 6 months.
  Other Names: Surveys
Behavioral: Breath Test — Breath test performed at 3 month and 6 month visit.
Behavioral: Proactive Cell Phone Smoking Cessation Counseling — Participant receives 11 phone calls from study staff over a 6-month period.
  Arms: Group 1 - Phone Call Support
Behavioral: Text Message Smoking Cessation Support — Participants receive text messages for support about quitting smoking over a 6 month period.
  Arms: Group 2 - Text Messaging Support

SUMMARY:
The goal of this research study is to compare 2 different phone-based programs for quitting smoking for people with HIV/AIDS.

DETAILED DESCRIPTION:
If participant agrees to take part in this study, the following will be done at the first visit (called the Baseline Visit):

* The study staff will give participant advice about quitting smoking. Participant will then set a quit date, after which they will plan to not smoke anymore.
* Participant will receive a 10-week supply of nicotine patches and instructions on how to use them.
* Participant will complete questionnaires on a laptop computer about their smoking habits, how much tobacco they use, how many times they have tried to quit, how ready they are to quit, and how dependent they are on nicotine. The questionnaires will take about 30 minutes to complete.

Participant will then be assigned to 1 of 2 study groups. Participant will have a 1 in 5 (20%) chance of being assigned to Group 1, and a 4 in 5 (80%) chance of being assigned to Group 2.

If participant is in Group 1:

* Participant will receive a telephone number to a hotline for them to use to call and talk to someone about quitting. Participant can call the hotline anytime they need support in their effort to quit smoking.
* Participant will also receive 11 phone calls from the study staff over a 6-month period. During each call, participant will be given support to help them quit. Each call will last about 15 minutes.

If participant is in Group 2:

* Participant will receive text messages for support about quitting smoking. In the first week, participant will get about 20 text messages. Each week, participant will receive fewer text messages, until they get 1 message per week by week 4. Participant will then get 1 message each week after that through month 6.
* Participant will also receive another text message 1 time each week from the study staff asking if they have smoked within the past 24 hours. Participant will be asked to respond to this text message either by sending a text back to the study staff or calling the study staff. If the study staff does not receive participant's response they may receive a phone call from the staff asking about their smoking status over the past 24 hours.

Follow-Up Visits (Both Groups):

Three (3) and 6 months after the Baseline Visit, you will complete questionnaires on a laptop computer and participant will be asked for more information about their smoking status. At this visit, participant will also be asked to blow into a cardboard tube to check for byproducts of smoking. These visits will last about 20 minutes each.

Length of Study:

Participant will be on study for about 6 months.

This is an investigational study.

Up to 1000 patients will take part in this study. All will be enrolled at Legacy Community Health Services Clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Receiving care for HIV/AIDS at a Legacy Community Health Services Clinic
2. 18 years of age or older
3. Self-reported current smoker (smoked at least 100 cigarettes in lifetime and smoking every day or most days)
4. Able to provide written informed consent to participate
5. English or Spanish speaking

Exclusion Criteria:

1. Positive history of a medical condition that precludes use of the nicotine patch
2. Current use of nicotine replacement therapy (NRT)
3. Current use of other smoking cessation medications (e.g., Chantix or Zyban)
4. Pregnant or nursing
5. Enrolled in another smoking cessation study
6. Unwilling to set a target quit date

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Smoking Abstinence | 3 months
  Smoking abstinence defined as biochemically confirmed 7-day abstinence. Expired CO will be used to biochemically verify abstinence.

CONTACTS AND LOCATIONS:
Overall Officials: Damon Vidrine, MS, DRPH, BA, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org